CLINICAL TRIAL: NCT06509191
Title: Effect of Melatonin Versus Placebo for Prevention of Delirium Among Medically Hospitalized Patients: Study Protocol for a Single-Center, Double-Blinded, Randomised Controlled Trial
Brief Title: The Use of Melatonin for Delirium Prevention in Medically Hospitalized Patients
Acronym: RESTORE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Dr. Abdullah Al Alawi, Sr. Consultant, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sultan Qaboos University
Record Dates: First submitted 2024-07-10; First posted 2024-07-19 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Delirium
Keywords: delirium; melatonin; Hospitalized; Medical
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Intervention Model Description: The study will be a randomized, double-blind, and parallel arm placebo-controlled trial which will take place at Sultan Qaboos University Hospital. All patients aged 65 years and over admitted through emergency department to General Internal Medical Units will be screen for eligibility.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Melatonin 5mg/day (Experimental): Intervention group 1: Melatonin 5mg/day
  * Study drug will be given at 20:00 - 22:00 daily, starting on the day of enrolment until discharge, death, or up to 5 days as most medically hospitalised patients at great risk of delirium in the first few days of admission.(20)
  * The study medication will be given by mouth or if needed, via the feeding tube followed by a flush with 20mL water.
  Interventions: Drug: Intervention 1
- Melatonin 8 mg/day (Experimental): Intervention group 2:Study drug will be given at 20:00 - 22:00 daily, starting on the day of enrolment until discharge, death, or up to 5 days as most medically hospitalised patients at great risk of delirium in the first few days of admission.(20)
  • The study medication will be given by mouth or if needed, via the feeding tube followed by a flush with 20mL water.
  Interventions: Drug: Intervention 2
- Placebo (Placebo Comparator): * Study drug will be given at 20:00 - 22:00 daily, starting on the day of enrolment until discharge, death, or up to 5 days as most medically hospitalised patients at great risk of delirium in the first few days of admission. (20)
  * The study medication will be given by mouth or if needed, via the feeding tube followed by a flush with 20mL water.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Intervention 1 — Melatonin 5mg/day
  Arms: Melatonin 5mg/day
Drug: Intervention 2 — Melatonin 8 mg/day
  Arms: Melatonin 8 mg/day
Other: Control — Placebo
  Arms: Placebo

SUMMARY:
The high prevalence of delirium in hospitalized older adults, with significant associated morbidity and mortality, emphasize the need for effective prevention strategies. Limited trials have explored melatonin's potential in preventing delirium among patients admitted to general medical wards. Previous trials on melatonin's preventive role in medical wards had limitations, necessitating a robust, double-blinded, placebo-controlled design with a larger sample size. This randomized, double-blind study of melatonin versus placebo aims to investigate the efficacy of melatonin, a neurohormone regulating the sleep-wake cycle, in preventing delirium among medically hospitalized patients aged 65 or older. Given the high prevalence of delirium in this population and its association with adverse outcomes, the study seeks to contribute valuable insights into an effective preventive strategy.

DETAILED DESCRIPTION:
Background and rationale:

Delirium, a neuropsychiatric syndrome, manifests acutely with altered consciousness, cognitive impairment, and inattention, showing a fluctuating course.1 Delirium can present as hyperactive, hypoactive, or mixed, posing challenges for identification, especially in the elderly.1 Recent systematic reviews reveal its presence in approximately 50% of hospitalized individuals aged 65 or older, with 15-25% developing delirium post major elective surgeries and up to 80% in intensive care units requiring mechanical ventilatory support.2 3 Various modifiable and non-modifiable risk factors contribute to delirium, emphasizing the need for appropriate interventions to reduce risk. 2 3 The presence of delirium in the elderly has been associated with poor health outcomes. A meta-analysis demonstrated a significant association with increased mortality risk at a 22-month follow-up (hazard ratio of 1.95).4 Unlike several other medical conditions, delirium-associated mortality has not declined over the past three decades. 5 Delirium is linked to higher mortality rates both during and after hospital admission, especially in critically ill patients with severe symptoms.6 It often results in prolonged hospital stays, including prolonged stay in the ICU, due to the condition's complexity and severity.7 Delirium is significantly associated with long-term cognitive impairment and an increased risk of dementia, with cognitive decline persisting beyond the hospital stay.7 8 It can also lead to poor functional recovery, affecting patients' ability to return to their previous level of independence and quality of life.6 The condition is associated with higher healthcare costs due to longer stays, increased need for specialized care, and potential readmissions. Additionally, patients experiencing delirium are more likely to be discharged to long-term care facilities rather than returning home, reflecting the impact on their functional and cognitive abilities.9 Non-pharmacological interventions are vital for preventing delirium in hospitalized patients, as treatment options for established delirium are limited. 10 These interventions focus on altering environmental and care practices to reduce delirium incidence. Multicomponent strategies, which include cognitive stimulation, sleep hygiene, re-orientation with familiar objects, and nutritional attention, significantly reduce delirium compared to standard care. Involving family members in patient care fosters patient-centered care and lowers delirium rates.11 Environmental modifications, such as reducing sensory deprivation and ensuring proper lighting, create a more familiar environment to prevent delirium.10 Cognitive and sensory stimulation help maintain orientation and cognitive function. Sleep hygiene and exercise programs support restful sleep and physical activity, respectively, aiding in delirium prevention.11 Despite extensive pharmacological interventions, no definitive advantages have emerged. Haloperidol, a prototypical first-generation antipsychotic, has been thoroughly studied for delirium treatment, yet the evidence supporting its efficacy remains limited. 12 Its administration failed to demonstrate significant advantages concerning delirium incidence, mortality, or length of hospital stay compared to a placebo.12 While olanzapine and quetiapine are potential pharmacological alternatives, their association with adverse events, including metabolic abnormalities and corrected QT (QTc) interval prolongation, raises concerns. Both drugs share similar risks for diabetes and cardiovascular events, but quetiapine may pose a higher risk for hyperlipidemia and ischemic stroke in certain populations.13 Olanzapine is more associated with weight gain.13 Due to this risk profile and a lack of substantial evidence supporting their effectiveness in preventing or treating delirium, these second-generation antipsychotics have not gained widespread clinical adoption.. 14 Although an altered sleep-wake cycle is not a diagnostic criterion for delirium, sleep deprivation and delirium share many epidemiologic, biochemical, and anatomic similarities.15 Nearly 75% of patients with delirium have sleep disorders, and the quality of sleep is an integral part of certain delirium screening tools.16 The diagnostic criteria for delirium, propsed by Trzepacz, Meagher, and Franco (TMF) Research Diagnostic Criteria, emphasize core domains including cognition, higher-level thinking, and circadian rhythm. These are evidenced by impaired attention (Criterion B), deficits in cognitive domains and disorganized thinking (Criterion C), and circadian disruptions such as sleep-wake cycle disturbances or motor activity changes (Criterion D). This framework provides a comprehensive basis for understanding delirium and its associations with sleep-wake cycle disruptions.17 Hence, the hypothesis emerges that preventing or treating sleep abnormalities could impact delirium. Melatonin, a neurohormone principally produced by the pineal gland at night, improves the quality of sleep and has hypnotic effects when administered exogenously. Studies have shown that melatonin circadian rhythm is disturbed in patients with delirium. 16 Melatonin improves sleep quality at doses ranging from 0.3 mg to 5 mg, with the optimal dose varying based on individual factors like age and health status.18 Higher doses may be beneficial for older adults and specific conditions such as postoperative recovery. Doses above 0.5 mg/day help in resetting the sleep-wake cycle.19 20 Melatonin also acts as an antioxidant, similar to glutathione and tocopherol, by scavenging hydroxyl and neutralizing peroxyl radicals, reducing cellular damage. 21 Due to its antioxidant properties, melatonin may offer neuroprotective effects and potentially diminish the risk of neurodegenerative diseases. 21 Utilizing melatonin in delirium treatment could thus address circadian rhythm disturbances and impact various hypothesized pathways in delirium development.

A systematic review and meta-analysis assessed the prophylactic effect of melatonin receptor agonists (MMRAs) on postoperative delirium (POD) in elderly patients. 22 Analyzing 11 randomized controlled trials with a total of 1,558 patients, the results revealed that the MMRA group had a significantly lower occurrence of postoperative delirium (POD) compared to the placebo group (risk ratio = 0.70, 95% confidence interval: 0.51-0.97, P < 0.05, I² = 59%). Due to high heterogeneity, a subgroup analysis was performed, which indicated that melatonin significantly reduced POD occurrence, supported by moderate-quality evidence, whereas ramelteon and tryptophan showed no significant impact.22 Another systematic review and meta-analysis was done to determine the preventive effect of melatonin on delirium in the intensive care unit, including six RCTs (n=2374 patients). 23 A meta-analysis of six studies involving 2,374 patients examined the effects of melatonin on delirium in intensive care settings. 23 Overall, melatonin did not significantly reduce the incidence of delirium in ICU patients (odds ratio [OR]: 0.71; 95% confidence interval [CI]: 0.46 to 1.12; p = 0.14), with notable heterogeneity among studies (I² = 74%). However, subgroup analysis revealed that melatonin significantly reduced delirium incidence in cardiovascular care unit (CCU) patients (OR: 0.52; 95% CI: 0.37 to 0.73; p = 0.0001), but not in general ICU (GICU) patients (OR: 1.14; 95% CI: 0.86 to 1.50; p = 0.35). Secondary outcomes showed no significant differences in all-cause mortality (OR: 0.85; 95% CI: 0.66 to 1.09; p = 0.20), length of ICU stay (mean difference [MD]: 0.33; 95% CI: -0.53 to 1.18; p = 0.45), or length of hospital stay (MD: 0.51; 95% CI: -1.17 to 2.19; p = 0.55) between the melatonin and placebo groups. 23

A recent systematic review and meta-analysis included three RCTs and six observational studies (n = 1211). All three RCTs compared melatonin to placebo, while most observational studies compared melatonin or ramelteon to antipsychotics. 24 Two RCTs reported the duration of delirium, showing a statistically significant reduction with melatonin compared to placebo (-1.72 days, 95% CI -2.66 to -0.77, p = 0.0004). Five observational studies examined the duration of delirium, but only one showed a significant reduction with ramelteon combined with antipsychotics compared to antipsychotics alone (6.6±1 vs. 9.9±1.3 days, p=0.048). Delirium severity showed mixed results; melatonin improved the BPRS score in one RCT, while other studies found no benefit. 24 In a randomized controlled trial comprising 497 patients admitted with acute decompensated heart failure, the administration of melatonin at a dosage of 3 mg/day for a duration of 7 days demonstrated a significant reduction in the incidence of delirium within the melatonin group compared to the placebo group (27.0% vs. 36.9%, P = 0.021). Safety assessments revealed comparable occurrences of rhabdomyolysis and abnormal hepatic function in both groups. 25 Most trials assessing the role of melatonin in preventing delirium were conducted in intensive care settings or surgical wards. There are very few trials involving hospitalized patients in medical wards. Another randomized clinical trial involving hospitalized individuals aged 65 or older (n=36 received melatonin, 33 received placebo) administered 3 mg of melatonin. The study concluded that the nightly use of 3 mg melatonin did not reduce the incidence of delirium. 29 Overall, the trial conducted on hospitalized patients in medical wards had limitations, including small sample sizes, variations in medication doses, and a lack of assessment of healthcare outcomes such as mortality, length of hospital stay, and hospital readmission associated with delirium. 29 The high prevalence of delirium in hospitalized older adults, with significant associated morbidity and mortality, highlights the need for effective prevention strategies. Despite extensive exploration of pharmacological interventions, current evidence lacks definitive advantages, and widely used antipsychotics present concerns. Recognizing the link between sleep disturbances and delirium, melatonin, a neurohormone regulating the sleep-wake cycle, emerges as a promising medication. Previous studies demonstrated mixed results, with some indicating a prophylactic effect on postoperative delirium, while others show no significant impact on delirium incidence in intensive care units. Importantly, limited trials have explored melatonin's potential in preventing delirium among patients admitted to general medical wards. Previous trials faced limitations such as small sample sizes and the use of very small doses of melatonin.

Objectives:

This study aims to investigate the efficacy of melatonin, a neurohormone regulating the sleep-wake cycle, in preventing delirium among medically hospitalized patients aged 65 years or older. Given the high prevalence of delirium in this population and its association with adverse outcomes, the study seeks to contribute valuable insights into an effective preventive strategy. The planned trial will be novel in focusing on patients admitted to general medical wards where evidence is scarce. It will utilize two doses of melatonin versus placebo and include a larger sample size to ensure good statistical power. This study's robust, double-blinded, placebo-controlled design will address the existing gaps and limitations, offering new insights into melatonin's preventive role against delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 65 years and above acutely admitted under the care of General Internal Medicine Unit

Exclusion Criteria:

* Patients admitted to the ward, however meeting requirement for vasopressors or non-invasive ventilation.
* Patient admitted through emergency to Intensive Care Unit (ICU) or High Dependency Unit (HDU).
* Aphasic patients.
* Patients with language barriers.
* Already taking melatonin or ramelteon at the time of randomization.
* Presence of delirium at the time of randomization.
* If enteral medications are contraindicated due to gastrointestinal conditions.
* If enteral medications are not allowed due to unavailability of nasogastric tube
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) (liver function tests) > 3 times the upper limit of normal.
* Patient on strong cytochrome P450 1A2 (CYP1A2) inhibitors (namely: fluvoxamine and viloxazine) .
* Patient with active alcohol drinking or admitted with alcohol withdrawal syndrome.
* Subject or proxy unable to provide informed consent within 24 hours of admission.
* Patients with the following autoimmune diseases (Rheumatoid arthritis, inflammatory bowel disease and systemic lupus erythematosus).
* Allergy to melatonin.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium | 5 days
  Incidence of delirium development during hospitalisation using the 3-Minute Diagnostic Confusion Assessment Method (3D-CAM).

SECONDARY OUTCOMES:
Onset time of delirium | 5 days
  The time from hospital admission to the first diagnosis of delirium is measured in hours or days from admission and is assessed daily during the first 5 days of hospitalization. The development of deleiriun will be ascertain assessed daily by trained research assessors, using the 3D-CAM tool.
Duration of delirium during hospitalization | 5 days
  The total time a patient remains in a state of delirium during the hospital stay is recorded in hours or days using the 3-Minute Diagnostic Confusion Assessment Method (3D-CAM). This duration is assessed daily during the first 5 days of hospitalization.
Sleep pattern and night awakenings | 5 days
  The quality of sleep, including the number of awakenings and disruptions during the night, is assessed using patient self-reports, nursing records, or information from attendants. Night awakenings are quantified by the number of instances per night and are evaluated nightly during the first 5 days of hospitalization by trained research assitant .
Days utilizing physical restraints. | 5 days
  The number of days physical restraints were used during hospitalization is recorded in days based on hospital records and staff documentation, and is assessed for first 5 days .
• Number of rescue medications during hospitalization. | 5 days
  The number of rescue medications, such as antipsychotics, administered for managing delirium symptoms is recorded.This is assessed during the first 5 days of hospitalization.
Length of hospital stay (LOS). | entire hospitalization period (up to 24 weeks)
  The total duration of hospitalization, from admission to discharge, is recorded in days and assessed at the end of the hospitalization.
Requirement to transfer to high dependency unit (HDU) or ICU | entire hospitalization period (up to 24 weeks)
  Whether the patient required transfer to HDU or ICU during hospitalization is recorded as a binary variable (yes/no), with reasons for transfer documented. This is assessed continuously during the hospitalization.
Inpatient all-cause mortality. | entire hospitalization period (up to 24 weeks)
  Inpatient all-cause mortality :Mortality occurring during the hospital stay, regardless of cause, is recorded as a binary variable (yes/no) from hospital records and is assessed for the entire hospitalization period.
28- day all-cause mortality | within 28 days post-discharge
  Mortality occurring within 28 days of hospital admission, regardless of cause, is recorded as a binary variable (yes/no) from follow-up records and is assessed within 28 days post-discharge
28- day all-cause mortality | 28 days post-discharge.
  Whether the patient was readmitted to the hospital within 28 days of discharge is recorded as a binary variable (yes/no) based on follow-up records, and is assessed within 28 days post-discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Oman

IPD SHARING:
Plan to Share IPD: Yes
The de-identified IPD will be made available to researchers upon reasonable request. Interested researchers should contact the study PI alalawi2@squ.edu.om and provide a brief proposal detailing the intended use of the data. Requests will be reviewed by the primary research team, and access will be granted following approval. Data will be shared through a secure data-sharing platform.
Supporting Information: Study Protocol
Time Frame: upon completion of the data analysis
Access Criteria: The de-identified IPD will be made available to researchers upon reasonable request

REFERENCES:
- [Background] Riviere J, van der Mast RC, Vandenberghe J, Van Den Eede F. Efficacy and Tolerability of Atypical Antipsychotics in the Treatment of Delirium: A Systematic Review of the Literature. Psychosomatics. 2019 Jan-Feb;60(1):18-26. doi: 10.1016/j.psym.2018.05.011. Epub 2018 May 31. PMID 30181002
- [Background] Shen YZ, Peng K, Zhang J, Meng XW, Ji FH. Effects of Haloperidol on Delirium in Adult Patients: A Systematic Review and Meta-Analysis. Med Princ Pract. 2018;27(3):250-259. doi: 10.1159/000488243. Epub 2018 Mar 8. PMID 29518791
- [Background] Burton JK, Craig LE, Yong SQ, Siddiqi N, Teale EA, Woodhouse R, Barugh AJ, Shepherd AM, Brunton A, Freeman SC, Sutton AJ, Quinn TJ. Non-pharmacological interventions for preventing delirium in hospitalised non-ICU patients. Cochrane Database Syst Rev. 2021 Jul 19;7(7):CD013307. doi: 10.1002/14651858.CD013307.pub2. PMID 34280303
- [Background] Al Huraizi AR, Al-Maqbali JS, Al Farsi RS, Al Zeedy K, Al-Saadi T, Al-Hamadani N, Al Alawi AM. Delirium and Its Association with Short- and Long-Term Health Outcomes in Medically Admitted Patients: A Prospective Study. J Clin Med. 2023 Aug 17;12(16):5346. doi: 10.3390/jcm12165346. PMID 37629388
- [Background] Goldberg TE, Chen C, Wang Y, Jung E, Swanson A, Ing C, Garcia PS, Whittington RA, Moitra V. Association of Delirium With Long-term Cognitive Decline: A Meta-analysis. JAMA Neurol. 2020 Nov 1;77(11):1373-1381. doi: 10.1001/jamaneurol.2020.2273. PMID 32658246
- [Background] Lozano-Vicario L, Garcia-Hermoso A, Cedeno-Veloz BA, Fernandez-Irigoyen J, Santamaria E, Romero-Ortuno R, Zambom-Ferraresi F, Saez de Asteasu ML, Munoz-Vazquez AJ, Izquierdo M, Martinez-Velilla N. Biomarkers of delirium risk in older adults: a systematic review and meta-analysis. Front Aging Neurosci. 2023 May 12;15:1174644. doi: 10.3389/fnagi.2023.1174644. eCollection 2023. PMID 37251808
- [Background] Wang CG, Qin YF, Wan X, Song LC, Li ZJ, Li H. Incidence and risk factors of postoperative delirium in the elderly patients with hip fracture. J Orthop Surg Res. 2018 Jul 27;13(1):186. doi: 10.1186/s13018-018-0897-8. PMID 30049276
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Chin YC, Koh GC, Tay YK, Tan CH, Merchant RA. Underdiagnosis of delirium on admission and prediction of patients who will develop delirium during their inpatient stay: a pilot study. Singapore Med J. 2016 Jan;57(1):18-21. doi: 10.11622/smedj.2016007. PMID 26831312
- [Derived] Al Alawi AM, Al Busaidi S, Al Rasbi SK, Al Farsi RS, Al Zeedy K, Al Huraizi AR, Al-Maqbali JS. Effect of melatonin versus placebo for the prevention of delirium among medically hospitalised older patients: a double-blinded randomised controlled trial (project RESTORE). BMJ Open. 2026 Jan 27;16(1):e107775. doi: 10.1136/bmjopen-2025-107775. PMID 41592826
- [Derived] Al-Maqbali JS, Al-Busaidi S, Al Farsi RS, Al Rasbi S, Al Zeedy K, Al Huraizi AR, Al Alawi AM. Effect of melatonin versus placebo for prevention of delirium among medically hospitalised patients: study protocol for a single-centre, double-blinded, randomised controlled trial (project RESTORE). BMJ Open. 2025 Feb 25;15(2):e094195. doi: 10.1136/bmjopen-2024-094195. PMID 40000080